CLINICAL TRIAL: NCT04599036
Title: Myoelectrolytically Controlled Device in Acute Rehabilitation After Stroke
Brief Title: EMG Controlled Device in Acute Rehabilitation After Acute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B3554-M
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Feasibility (Experimental): To explore if the feasibility of adding an EMG controlled device to the acute rehabilitation for stroke subjects with severe arm deficit.
  Interventions: Device: MARK

INTERVENTIONS:
Device: MARK — EMG controlled arm orthosis

SUMMARY:
Stroke is a medically relevant problem for the aging population. Individuals with stroke experience a high amount of arm functional deficits despite receiving rehabilitation. Functional deficits can be improved by combining rehabilitation with innovative rehabilitative tools that target the brain mechanisms that guide the recovery early after stroke. This study aims to explore the feasibility of implementing an EMG controlled device in the acute rehabilitation for stroke survivors with severe arm deficit. This study will determine if adding such a technology improve the clinical outcomes for subjects with severe arm impairments beyond the levels achieved by standard care in attempt to increase their chances to independently perform activities of daily living.

DETAILED DESCRIPTION:
During the first weeks after the onset of stroke, the injured brain undergoes several neural mechanisms, a process known as neuroplasticity, that intend to reorganize the neural connectivity and repair the damaged tissue around the injury region. Several studies revealed that rehabilitation during this acute period of injury would enhance the functional outcome of the paretic arm presumably by modulating the heightened neuroplastic mechanism. Specifically, it has been suggested that novel interventions that interact with the neuroplastic mechanisms of recovery are particularly needed for stroke survivors whom initial arm impairments are severe.

The rationale of this study is to explore if an EMG controlled device can be added to the acute rehabilitation for stroke subjects with severe arm deficit. The study will also investigate if the application of such a device would lead to an even better enhancement of clinical outcomes compared to standard care. Because of such neurophysiological changes during the acute phase, the study aims to correlate the neurophysiological changes with the enhancement gained as a result of practicing with an EMG controlled device in this population. Thus, test the premise that adding practice with an EMG controlled device to the acute rehabilitation of subjects with severe arm impairments acts as novel rehabilitative tool that interact with the neuroplastic mechanisms of recovery to enhance clinical outcomes for these subjects.

ELIGIBILITY:
Inclusion Criteria:

* Veterans over 18 years of age
* 2 days to 6 months since the onset of ischemic stroke
* Adequate range of motion at the elbow, forearm, wrist, and hand to wear the device.
* Ability to generate volitional, consistent, and detectable EMG signals from the upper arm and forearm sensor sites with wrist in neutral or flexed positions as detected by the Myopro software
* MAS score 3 for the biceps, triceps, supinators and pronators of the impaired arm
* Able to read and comprehend the English language
* Able to follow directions
* Medically and psychologically stable.

Healthy Controls:

Over 18 years of age No history of neurological or muscular problems that affect arm function

Exclusion Criteria:

Hemorrhagic stroke

* Previous strokes affecting motor function on the opposite side.
* Fugl-Meyer score of 2 on the following 3 items:

  1) finger mass extension, 2) grasp #1 test, and 3) shoulder flexion 90 - 180 degrees, elbow at 0 degree, and forearm neutral.
* Shoulder subluxation, pain or dislocation
* Shoulder passive range of motion < 45 degrees in flexion and abduction
* Fixed upper limb contractures on the impaired arm and hand
* Unable to safely support the weight of their arm plus 4 lbs (1.82 kg; the weight of the device) without pain even with arm supported.
* Skin rash or open wound on impaired arm
* Involuntary movements of the impaired arm
* Pacemaker or other implanted devices
* Metal in the skull
* Claustrophobia, or inability to operate the MRI patient call button
* Past history of seizures
* Family history of medication refractory epilepsy
* Chronic sleep deprivation, ongoing untreated sleep disorder
* Pregnancy or pregnancy planning during the study period
* Currently taking medications or substances that lower the threshold for onset of seizure.
* Inability to understand English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-07 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in arm impairment using Fugl-Meyer assessment (FMA) | Change from Baseline arm impairment after 6 weeks
  Measure of arm impairment. Scores on the FMA may range from 0-66 points, with higher score indicating better performance.

SECONDARY OUTCOMES:
Changes in arm function using Action Research Arm Test (ARAT) | Change from Baseline arm function after 6 weeks
  Measure of arm function. Scores on the ARAT may range from 0-57 points, with higher score indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ahlam Salameh, PhD MSc, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No